CLINICAL TRIAL: NCT04556604
Title: Consent for Surgery During the COVID-19 Pandemic
Brief Title: Surgical Consent During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Medway Primary Care Trust (Other Government)
Responsible Party: Principal Investigator, Oloruntobi Rotimi, Dr, Medway Primary Care Trust
Other Study IDs: 2021.016N
Record Dates: First submitted 2020-09-18; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Consent

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: First cycle of the audit on consenting practice pre intervention
- 2: Second cycle of the audit on consenting practice to assess change following intervention
  Interventions: Behavioral: Educational meetings and visual prompts
- 3: Third cycle of the audit on consenting practice to assess long term compliance
  Interventions: Behavioral: Educational meetings and visual prompts

INTERVENTIONS:
Behavioral: Educational meetings and visual prompts — Information was disseminated to trainees via informal meeting or dedicated audit meetings with the aid of visual prompts
  Groups: 2; 3

SUMMARY:
Multiloop audit of consenting practice in surgical procedures during the COVID-19 pandemic

ELIGIBILITY:
Exclusion Criteria:

* Children (under 18 years old)
* Participants who lack capacity and therefore cannot be consented appropriately

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults presenting with general surgical, vascular or breast surgical issues that require surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Compliance to consenting practice | 3 months
  The number of patients being consented for COVID-19 infection in the lead up to surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Medway NHS Foundation Trust, Gillingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
On request, IPD may be shared. This will include anonymised data collected during the study period